CLINICAL TRIAL: NCT06456879
Title: Clinical Performance and Convenience of Three Types of Crowns as Esthetic Alternatives to Stainless Steel Crowns for Primary Molars
Brief Title: Clinical Performance and Convenience of Four Types of Crowns for Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M01010222
Record Dates: First submitted 2024-05-19; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-03

CONDITIONS: Crown of Tooth With Poor Contour
Keywords: crowns; molars; wear; zirconia; hybrid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stainless Steel Crown (Active Comparator): crown
  Interventions: Other: extra-coronal restoration type
- • NuSmile zirconia crown (Active Comparator): crown
  Interventions: Other: extra-coronal restoration type
- • CAD CAM zirconia crown (Active Comparator): crown
  Interventions: Other: extra-coronal restoration type
- • CAD CAM hybrid crown (Active Comparator): crown
  Interventions: Other: extra-coronal restoration type

INTERVENTIONS:
Other: extra-coronal restoration type — primary molar crown type

SUMMARY:
This study will be conducted to assess the clinical performance and convenience of three types of crowns as esthetic alternatives to stainless steel crown for primary molars:

* The prefabricated commercially available zirconia crowns (NuSmile®) (NZC).
* The locally manufactured zirconia crowns created via Computer-Aided Design/Computer-Aided Manufacturing (CAD/CAM) system (CCZC).
* The locally manufactured hybrid ceramic crowns created via Computer-Aided Design/Computer-Aided Manufacturing (CAD/CAM) system (CCHC).

DETAILED DESCRIPTION:
Eighty lower second primary molars will be divided into 4 groups:

* Group 1(n=20): receive 3M™ ESPE™ Stainless Steel crowns for Primary Molars.
* Group 2 (n=20): receive the prefabricated commercially available zirconia crowns (NuSmile®) (NZC).
* Group 3 (n=20): receive the locally manufactured zirconia crowns created via (CAD/CAM) system (CCZC).
* Group 4 (n=20): receive the locally manufactured hybrid ceramic crowns created via (CAD/CAM) system (CCHC).

Clinical and radiographic examination of the primary molar will be conducted to ensure compliance with the study criteria. Oral health instructions will be given to the child and parents then the application of local anesthesia.

1. Stainless steel crowns:

   Reduction of occlusal surface by about 1.5 mm using a flame shaped diamond bur to produce a uniform occlusal reduction. Proximal reduction using a long and tapered diamond bur to allow the probe to pass through the contact area. An appropriate size will be selected according to mesiodistal width of the prepared tooth and a trial fit will be carried out before cementation. The crown should remain no more than 1 mm subgingivally.(21)
2. Zirconia and hybrid ceramic crowns:

   The appropriate size of the posterior crown will be selected for the tooth chosen for treatment. The occlusal surface will be reduced by 1-2 mm by using a flame bur after evaluation of the occlusal relationships. The interproximal areas will be opened followed by reduction of the crown dimensions by 0.5-1.25 mm using a tapered diamond bur making the contour of the prepared tooth consistent with the natural contour. The prepared tooth walls will be finished with a 1-2 mm subgingival feather-edge preparation using a thinner pointed tapered diamond bur.

   The selected crown will be tested for appropriate fit before the final cementation. Finally, the prepared tooth will be cleaned from saliva, blood, and the remnants of preparation and ready for cementation.(15) The selected crown will be cleaned and then filled with resin modified glass ionomer cement. The crown will be applied with no resistance to the fully seated position on the tooth (Passive Fit) since forcing the crown to place can produce micro-fractures in the zirconia structure. Excess cement will be removed using a dental probe and dental floss.

   Clinical evaluation:

   o Evaluation criteria concerning the clinical performance are

1) The Gingival Index (GI)(22) will be measured by the William Gingival Probe with a blunt-ended instrument gently placed within the gingival gutter around each tooth to be crowned/previously crowned, and the values will be as follows: 0 = normal gingiva

1. = mild inflammation: a slight change in color, slight edema, no bleeding on probing
2. = moderate inflammation: redness, edema, and glazing, or bleeding on probing
3. =severe inflammation: marked redness and edema, a tendency toward spontaneous bleeding, ulceration.

2) Plaque Index (PI)(22) will be measured by passing the gingival probe around each tooth to be crowned/previously crowned, and the values will be as follows: 0 = no plaque

1= film at the gingival margin and adjacent tooth 2 = moderate accumulation of plaque 3 = abundance of plaque.

Crown retention (23) will be measured as follows:

0 = present.

1 = absent.

Crown integrity(24) will be measured as follows:

0 = intact.

1. = crack present.
2. = fracture present.
3. = crown lost.

Marginal adaptation will be measured clinically and radiographically:

1) All crowns will be evaluated clinically at baseline, 3rd, 6th, 9th and 12th months and scored as follows:(25) 0 = Margin not discernible, probe does not catch.

1. = Probe catches on margin but no gap on probing.
2. = Probe catches on margin and a gap on probing.
3. = Crown fractured or missing. 2) All crowns will be evaluated radiographically at baseline, 6th, and 12th months to check the marginal adaptation.

Color stability(26) will be measured as follows:

0 = Unchanged.

1 = Minor deviation from original. Wear of the antagonistic natural enamel. To evaluate the wear of the antagonistic natural enamel of primary molar, a rubber base impressions will be made immediately (baseline) and at 1 year after cementation. The resulting casts will be scanned (using a 3D scanner), and 3D softare will be used to calculate the maximum amount of linear wear. (27)

o Evaluation criteria regarding the crown convenience: Time elapsed since the start of tooth preparation till the crown cementation. Anxiety using the Facial Image Scale (FIS).(28) The Facial image scale comprises a row of five faces ranging from very happy to very unhappy. The children were asked to point at which face they felt most like at that moment. The scale is scored by giving a value of one to the most positive affect face and five to the most negative affect face. Facial Image Scale has a fixed number of faces (not a continuous line) for the children to choose from, thus making it easier to score in a clinical situation, and easier for very young children to understand.

ELIGIBILITY:
Inclusion Criteria:

* Children between 4-8 years old.
* Definitely positive or positive behavior according to Frankl behavior rating scale.
* The lower second primary molar with one or more indications for crown restoration.

Exclusion Criteria:

* The child does not have occlusal problems or periodontal diseases
* The child does not take medications that lead to symptoms of periodontal diseases.

Ages: 4 Years to 8 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2022-02-05 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
the gingival index | 12 months
  0 = normal gingiva
  1. = mild inflammation
  2. = moderate inflammation
  3. = severe inflammation
Crown retention | 12 months
  0 = present.
  1 = absent.
Crown integrity | 12 months
  0 = intact.
  1. = crack present.
  2. = fracture present.
  3. = crown lost.
Color stability | 12 months
  0 = Unchanged.
  1. = Minor deviation from original.
  2. = Unacceptable discoloration.
Plaque Index | 12 months
  0 = no plaque
  1= film at the gingival margin and adjacent tooth 2 = moderate accumulation of plaque 3 = abundance of plaque.

SECONDARY OUTCOMES:
wear of opposing natural teeth. | 12 months
  To evaluate the wear of the antagonistic natural enamel of primary molar, the upper arch was scanned using an intraoral scanner immediately, (6 months and 1 year after cementation. Both 3d images were placed in the same position and compared using the CAD software to calculate the amount of linear wear on millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Diana M Amer, MASTER, Principal Investigator — Mansoura University; Abeer M Abdellatif, Phd, Study Chair — Mansoura University
Locations (2):
- Egypt (2):
  - Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahlia Governorate
  - Mansoura university, Al Mansurah, Dakahlya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amer DM, Abdellatif AM. In vivo evaluation of the enamel wear of primary molar against four types of crowns using the intra-oral scanner. BMC Oral Health. 2024 Nov 27;24(1):1438. doi: 10.1186/s12903-024-05206-5. PMID 39604941